CLINICAL TRIAL: NCT01585909
Title: Evaluation of Intestinal Brush Border Enzyme Function in Patients With SIRS and Septic Shock Compared to Control Patients
Brief Title: Evaluation of Intestinal Brush Border Enzyme Function in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Holzinger, MD, Assoc Prof, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BBM_septic_shock
Record Dates: First submitted 2012-04-12; First posted 2012-04-26 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Critical Illness; Septic Shock; SIRS
MeSH Terms: conditions — Critical Illness; Shock, Septic | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Septic Shock (Other): Activity of the brush border membrane enzymes intestinal alkaline phosphatase, maltase and lactase, as well as brush border morphology determined from duodenal biopsies in patients with septic shock
  Interventions: Procedure: Gastroscopy
- SIRS (Other): Activity of the brush border membrane enzymes intestinal alkaline phosphatase, maltase and lactase, as well as brush border morphology determined from duodenal biopsies in patients with SIRS
  Interventions: Procedure: Gastroscopy
- healthy/controls (Other): Activity of the brush border membrane enzymes intestinal alkaline phosphatase, maltase and lactase, as well as brush border morphology determined from duodenal biopsies in patients without SIRS/septic shock
  Interventions: Procedure: Gastroscopy

INTERVENTIONS:
Procedure: Gastroscopy — When gastroscopy is indicated for clinical reasons, duodenal biopsies to determine the activity of the brush border membrane enzymes intestinal alkaline phosphatase, maltase and lactase, as well as assessing brush border morphology are taken

SUMMARY:
The purpose of this study is to evaluate the role of several enzymes of the gut mucosa in preventing invasion of gastrointestinal bacteria.

DETAILED DESCRIPTION:
Systemic Inflammatory Response Syndrome (SIRS), sepsis, septic shock and concomitant multiorgan failure are major causes of morbidity and mortality in intensive care units. During SIRS and septic shock the role of the gut seems to be uncertain. As it serves as an intestinal barrier which allows the symbiotic relationship between man and enteric bacteria, increased gut permeability during critical illness is accused to promote sepsis. Brush border enzymes have the ability to detoxify lipopolysaccharides and prevent bacterial invasion across the gut mucosal barrier. A reduced brush border enzyme function could contribute to the gastrointestinal intolerance in critically ill patients, which is frequently observed. The aim of this study is to assess the influence of SIRS and septic shock on brush border enzyme morphology and function in men.

ELIGIBILITY:
Septic Shock:

Recruitment and inclusion criteria

* 15 mechanically ventilated critically ill patients fulfilling criteria of SIRS (2 symptoms: RR > 20/min, HR > 90/min, Temp. > 38°/< 36°, 12G/l< WBC < 4G/l; assumed or proven infection, persistent hypotension refractory to fluid therapy and need for vasopressors.
* Time window for inclusion: up to 72h after onset of symptoms

Exclusion criteria

* PLT < 50G/l,
* PT < 50%,
* Continuous therapeutic anticoagulation,
* DIC, st. p. MCI within 14 days,
* Gastrointestinal perforation,
* Age < 18 years,
* Age > 80 Years

SIRS:

Recruitment and inclusion criteria

* 15 mechanically ventilated critically ill patients fulfilling criteria of SIRS (2 symptoms: RR > 20/min, HR > 90/min, Temp. > 38°/< 36°, 12G/l < WBC < 4G/l; assumed or proven infection
* Time window for inclusion: up to 72h after onset of symptoms

Exclusion criteria:

* PLT < 50G/l,
* PT < 50%, continuous therapeutic anticoagulation,
* DIC, st. p. MCI within 14 days,
* Gastrointestinal perforation,
* Age < 18 years,
* Age > 80 Years

Healthy/controls:

* 15 control subjects will be recruited from the outpatient ward referred to the endoscopy of the Department of Medicine III - Division of Gastroenterology and Hepatology for upper GI-endoscopy because of epigastric pain or reflux symptoms.

Inclusion criteria:

* Signed informed consent

Exclusion criteria:

* Patients with diarrhea of unknown origin, IBD or known celiac disease
* Age < 18 years
* Age > 80 Years
* PLT < 50G/l, PT < 50%
* Therapeutic oral anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
activity of the brush border membrane enzyme intestinal alkaline phosphatase | at inclusion
  Duodenal biopsies will be taken on day 0 (at inclusion) and will be subsequently frozen. Determination of enzyme activity will be done within 28 days.

SECONDARY OUTCOMES:
activity of the brush border membrane enzyme maltase | at inclusion
  Duodenal biopsies will be taken on day 0 (at inclusion) and will be subsequently frozen. Determination of enzyme activity will be done within 28 days.
activity of the brush border membrane enzyme lactase | at inclusion
  Duodenal biopsies will be taken on day 0 (at inclusion) and will be subsequently frozen. Determination of enzyme activity will be done within 28 days.
Brush border morphology | at inclusion
  Duodenal biopsies will be taken on day 0 (at inclusion) and will be subsequently frozen. Determination of enzyme activity will be done within 28 days.
ICU mortality | at ICU discharge
  only for groups "septic shock" and "SIRS"
hospital mortality | at hospital discharge
  only for groups "septic shock" and "SIRS"
mortality (6 months) | 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria